CLINICAL TRIAL: NCT06936787
Title: A Prospective, Single-center, Open-label, Single Ascending Dose Study to Evaluate the Safety and Tolerability of Intravitreal Injection of IGT001 in Adult Patients With Retinitis Pigmentosa
Brief Title: An Open-label, Dose-ascending Study of IGT001 for Retinitis Pigmentosa
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Clinical Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INGEL-01
Record Dates: First submitted 2025-04-08; First posted 2025-04-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGT001 (Experimental)
  Interventions: Drug: IGT001

INTERVENTIONS:
Drug: IGT001 — Study drugs

SUMMARY:
This is an investigator-initiated, prospective, single-center, open-label, single ascending dose clinical study. The study aims to evaluate the safety, tolerability, and potential efficacy of intravitreal injection of IGT001 in patients with retinitis pigmentosa across different dose groups.

IGT001 is administered as a single intravitreal injection in the study eye under local anesthesia. Participants will be discharged on the day of treatment, provided that their visual acuity and intraocular pressure are close to baseline levels, and no clinically significant abnormalities in vital signs are observed compared to pre-injection values. The decision for discharge will be determined by the investigator's assessment.

DETAILED DESCRIPTION:
The study's dose groups are divided based on concentration into four cohorts: the low-concentration cohort (0.5 × 10⁶ hRP-50 µL), the medium-concentration cohort (1.0 × 10⁶ hRP-50 µL), the high-concentration cohort (2.0 × 10⁶ hRP-50 µL), and the target-concentration cohort.

Participants in the four cohorts will undergo a one-year follow-up as specified in the protocol. They will also be encouraged to participate in an additional one-year follow-up study to assess the long-term safety and tolerability of IGT001 after completing the main study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years at the time of signing the informed consent form, regardless of gender
* Clinical diagnosis of retinitis pigmentosa based on medical history and specialized examinations
* Willing to undergo genetic mutation testing, with results confirming known genetic mutations associated with hereditary retinal degeneration and related diseases
* Willing to provide blood samples for HLA typing
* Blood cell counts (hematocrit, hemoglobin, white blood cells, platelets) within the normal range, or outside the normal range but deemed clinically insignificant by the investigator
* Negative screening results for infectious diseases (hepatitis B, hepatitis C, and HIV), with no history of drug abuse (confirmed by negative urine test)
* Female participants of childbearing potential (defined as those who have not undergone surgical sterilization or have not been postmenopausal for at least one year) must undergo a urine pregnancy test at the time of admission (before injection), and the result must be negative.Female or male participants of childbearing potential must use medically approved contraceptive measures, such as abstinence, intrauterine devices (IUDs), or dual barrier methods (e.g., condom plus diaphragm), for at least 30 days before treatment and at least one year after treatment

Exclusion Criteria:

* As determined by the investigator, the study eye has concurrent conditions in addition to retinitis pigmentosa that:

  1. Affect central vision, or
  2. Increase the safety risk for the participant, or
  3. Impact efficacy or safety assessments or data collection, or
  4. Require surgical or medical intervention due to ocular diseases or history, such as retinal detachment or a history of retinal detachment, wet age-related macular degeneration, diabetic macular edema, retinal vein occlusion, uveitis, optic nerve disease, a history of glaucoma or ocular hypertension, severe or grade 3 non-proliferative diabetic retinopathy, proliferative diabetic retinopathy, significant media opacity, or an inability to achieve adequate pupil dilation
* The study eye cannot rule out the differential diagnosis of pseudoretinitis pigmentosa or cancer-associated retinopathies.
* History of malignant tumors (except for patients in remission for more than five years and those with basal cell carcinoma of the skin), end-stage major organ diseases (including heart failure, severe arrhythmias, stroke or transient ischemic attack, immunosuppressive or autoimmune conditions, severe mental disorders, epilepsy, chronic obstructive pulmonary disease, renal failure, or any chronic systemic disease requiring continuous systemic corticosteroids, anticoagulants, or immunosuppressive therapy)
* History of glaucoma in either eye or a glaucoma diagnosis at screening
* History of ocular hypertension in either eye or a diagnosis of ocular hypertension at screening
* Intraocular pressure (IOP) > 21 mmHg in either eye or current use of any intraocular pressure-lowering medications
* History of allergy, intolerance, or adverse reactions to any procedures involved in the study, including but not limited to a history of allergy/adverse reactions to contrast agents, needle phobia, or hemophobia
* History of ocular surface damage or drug-induced toxicity from medications such as deferoxamine, chloroquine/hydroxychloroquine (Plaquenil), tamoxifen, phenothiazines, or ethambutol
* History of allergy or adverse reactions to products containing dimethyl sulfoxide (DMSO)
* History of allergy to gentamicin
* Inability or unwillingness to comply with any study-related procedures, including genetic testing, blood sample collection, clinical examinations, or procedures requiring pupil dilation, topical anesthesia, or contrast agent injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
AE or SAE | 1 year
  The incidence of adverse events (AE) or serious adverse events (SAE)
The incidence of DLT | 28 days
  DLT

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No